CLINICAL TRIAL: NCT02913313
Title: Phase 1/2a First-In-Human Study of BMS-986207 Monoclonal Antibody Alone and in Combination With Nivolumab or With Nivolumab and Ipilimumab in Advanced Solid Tumors
Brief Title: A Study of BMS-986207 Given Alone and in Combination With Nivolumab or With Nivolumab and Ipilimumab in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA020-002; 2016-002263-34 (EudraCT Number)
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Results first posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Broad Solid Tumor
Keywords: First line NSCLC
MeSH Terms: interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1A: Dose Escalation Monotherapy (Experimental)
  Interventions: Drug: BMS-986207
- Part 1B: Dose Escalation Combination Therapy (Experimental)
  Interventions: Drug: BMS-986207; Biological: Nivolumab
- Part 2A: Expansion Monotherapy (Experimental)
  Interventions: Drug: BMS-986207
- Part 2B: Expansion Combination Therapy (Experimental)
  Interventions: Drug: BMS-986207; Biological: Nivolumab
- Part 1C: Triplet Cohort (Experimental)
  Interventions: Drug: BMS-986207; Biological: Nivolumab; Biological: Ipilimumab
- Part 2C: Triplet Expansion (Experimental)
  Interventions: Drug: BMS-986207; Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Drug: BMS-986207 — Specified dose on specified days
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
  Arms: Part 1B: Dose Escalation Combination Therapy; Part 1C: Triplet Cohort; Part 2B: Expansion Combination Therapy; Part 2C: Triplet Expansion
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy
  Arms: Part 1C: Triplet Cohort; Part 2C: Triplet Expansion

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of experimental medication BMS-986207 by itself, in combination with Nivolumab, and in combination with both nivolumab and ipilimumab in participants with solid cancers that are advanced or have spread.

ELIGIBILITY:
Inclusion Criteria:

* Must have pre-existing or prior programmed death-ligand 1 (PD-L1) immunohistochemistry (IHC) results within 3 months of enrollment from testing of tumor tissue; PD-L1 expression must be tumor cell positive ≥ 1% for a participant to be eligible for enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria; radiographic tumor assessment performed within 28 days before randomization

Exclusion Criteria:

* Primary central nervous system (CNS) disease, or tumors with CNS metastases as the only site of disease. Controlled brain metastases will be allowed to enroll
* Other active malignancy requiring concurrent intervention
* Uncontrolled or significant cardiovascular disease
* Active, known, or suspected autoimmune disease
* NSCLC without prior treatment in the advanced or metastatic setting (Part 2C)

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-11-30 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (6):
  - Local Institution - 0001, Hackensack, New Jersey
  - Local Institution - 0003, New York, New York
  - Local Institution - 0012, Philadelphia, Pennsylvania
  - Local Institution - 0002, Philadelphia, Pennsylvania
  - Local Institution - 0009, Pittsburgh, Pennsylvania
  - Local Institution - 0010, Salt Lake City, Utah
- Argentina (3):
  - Local Institution - 0023, CABA, Buenos Aires F.D.
  - Local Institution - 0019, Córdoba, Córdoba Province
  - Local Institution - 0022, Buenos Aires, Distrito Federal
- Local Institution - 0006, Nedlands, Western Australia, Australia
- Canada (2):
  - Local Institution - 0008, Ottawa, Ontario
  - Local Institution - 0007, Toronto, Ontario
- Local Institution - 0021, Santiago, Santiago Metropolitan, Chile
- Japan (2):
  - Local Institution - 0004, Kashiwa-shi, Chiba
  - Local Institution - 0005, Chuo-ku, Tokyo
- Romania (4):
  - Local Institution - 0017, Bucharest
  - Local Institution - 0016, Cluj-Napoca
  - Local Institution - 0018, Craiova
  - Local Institution - 0015, Florești
- Local Institution - 0020, Singapore, Singapore

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not randomized in Part 2B arm.
Groups:
- Part 1A BMS-986207 Safety Run In: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with total 48 mg of BMS-986207 as 60 minutes intravenous infusion in one cycle (each cycle of 8 weeks).
- Part 1A BMS-986207 20 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 20 milligram of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every 2 weeks (q2w).
- Part 1A BMS-986207 80 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 80 milligram of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every 2 weeks (q2w).
- Part 1A BMS-986207 240 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 240 milligram of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every 2 weeks (q2w).
- Part 1A BMS-986207 800 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 800 milligram of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every 2 weeks (q2w).
- Part 1A BMS-986207 1600 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 1600 milligram of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every 2 weeks (q2w) or 2 doses of BMS-986207 administered every 4 weeks (q4w).
- Part 2A BMS-986207 800 mg (CRC): Participants with colorectal cancer (CRC) were administered with 800 milligram of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every 2 weeks (q2w).
- Part 1B BMS-986207 80 mg + Nivolumab 240 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 80 mg of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every q2w. Participants were also administered with Nivolumab 240 mg as 60 minutes intravenous infusion for up to maximum of 6 cycles and each cycle comprise 4 doses of Nivolumab administered q2w.
- Part 1B BMS-986207 240 mg + Nivolumab 240 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 240 mg of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered every q2w. Participants were also administered with Nivolumab 240 mg as 60 minutes intravenous infusion for up to maximum of 6 cycles and each cycle comprise 4 doses of Nivolumab administered q2w.
- Part 1B BMS-986207 1600 mg + Nivolumab 480 mg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 1600 mg of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered q4w. Participants were also administered with Nivolumab 480 mg as 60 minutes intravenous infusion for up to maximum of 6 cycles and each cycle comprise 4 doses of Nivolumab administered q4w.
- Part 1B: BMS-986207 480 mg + Nivolumab 480 mg: Participants with CRC or ovarian cancer or hepatocellular carcinoma were administered with 480 mg of BMS-986207 as 60 minutes intravenous infusion for up to maximum of 6 cycles (each cycle is of 8 weeks). Each cycle comprise 4 doses of BMS-986207 administered q4w. Participants were also administered with Nivolumab 480 mg as 60 minutes intravenous infusion for up to maximum of 6 cycles and each cycle comprise 4 doses of Nivolumab administered q4w.
- Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 1600 mg of BMS-986207 every 3 weeks (q3w) as 60 minutes intravenous infusion for up to PD, unacceptable toxicity, or other protocol defined reasons or maximum of 2 years. Participants were also administered with Nivolumab 360 mg as 60 minutes intravenous infusion every 3 weeks (q3w) and Ipilimumab 1 mg/kg as intravenous infusion every 6 weeks at least 30 minutes after completion of the Nivolumab infusion.
- Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg: Participants with advanced solid tumors (metastatic, recurrent and/or unresectable) were administered with 600 mg of BMS-986207 every 3 weeks (q3w) as 60 minutes intravenous infusion for up to PD, unacceptable toxicity, or other protocol defined reasons or maximum of 2 years. Participants were also administered with nivolumab 360 mg as 60 minutes intravenous infusion every 3 weeks (q3w) and ipilimumab 1 mg/kg as intravenous infusion every 6 weeks at least 30 minutes after completion of the nivolumab infusion.
- Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg: Participants with first-line non-small cell lung cancer were administered with 600 mg of BMS-986207 every 3 weeks (q3w) as 60 minutes intravenous infusion for up to PD, unacceptable toxicity, or other protocol defined reasons or maximum of 2 years. Participants were also administered with nivolumab 360 mg as 60 minutes intravenous infusion every 3 weeks (q3w) and ipilimumab 1 mg/kg as intravenous infusion every 6 weeks at least 30 minutes after completion of the nivolumab infusion.
Period: Overall Study
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Started | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not Completed | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17 | 5
Not completed — DISEASE PROGRESSION | 1 | 2 | 2 | 4 | 6 | 4 | 19 | 3 | 4 | 4 | 11 | 5 | 14 | 3
Not completed — Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Other reasons | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — ADVERSE EVENT UNRELATED TO STUDY DRUG | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Not completed — STUDY DRUG TOXICITY | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Total
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5 | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 | 70.0 (2.83) | 61.0 (6.24) | 65.5 (12.61) | 56.4 (13.99) | 59.3 (9.43) | 60.1 (10.16) | 66.5 (3.11) | 48.8 (8.85) | 56.3 (19.57) | 63.9 (13.19) | 67.8 (10.03) | 56.9 (12.68) | 67.4 (8.91) | 60.7 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 4 | 2 | 9 | 3 | 1 | 2 | 4 | 3 | 9 | 1 | 45
  Male | 0 | 0 | 1 | 2 | 4 | 2 | 11 | 1 | 3 | 2 | 14 | 3 | 9 | 4 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 6
  Not Hispanic or Latino | 1 | 2 | 3 | 3 | 5 | 3 | 11 | 3 | 3 | 3 | 16 | 4 | 15 | 1 | 73
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 3 | 1 | 7 | 1 | 1 | 1 | 2 | 1 | 1 | 3 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 0 | 1 | 2 | 1 | 1 | 10 | 0 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 4
  White | 1 | 2 | 2 | 4 | 6 | 3 | 15 | 4 | 3 | 2 | 16 | 2 | 7 | 5 | 72
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. A Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization.
Time Frame: From first dose (Day 1) untill 100 days after last dose (Up to approximately 27 months)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
Participants
  Participants with any Adverse Events | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
  Participants with Serious Adverse Events | 1 | 0 | 3 | 3 | 5 | 1 | 11 | 3 | 2 | 1 | 6 | 4 | 11 | 5
  AEs leading to treatment discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 3

2. Primary Outcome: Number of Participants Who Died
Description: Participants who died with any cause are considered in the analysis.
Time Frame: From first dose (Day 1) untill 100 days after last dose (Up to approximately 27 months)
Population: All Treated Participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
Participants | 1 | 0 | 3 | 1 | 1 | 1 | 8 | 2 | 2 | 1 | 1 | 1 | 3 | 1

3. Primary Outcome: Part 1A, 1B and 1C and 2A: Number of Participants With Dose Limiting Toxicities
Description: Criteria for Dose-Limiting Toxicities (DLTs): Hepatic DLTs (excluding HCC): Grade (Gr) 4 elevations in AST, ALT, ALP, or total bilirubin. Gr 3 elevations in AST, ALT, or ALP >5 days, with symptoms, or bilirubin >2xULN without cholestasis. Gr 2 AST or ALT with symptomatic liver inflammation. AST or ALT >3xULN and bilirubin >2xULN without cholestasis. Hepatic DLTs for HCC: AST or ALT >10xULN for >2 weeks. AST or ALT >15xULN. Total bilirubin >8xULN (elevated at entry) or >5xULN (normal at entry). ALT ≥10xULN and bilirubin ≥2xULN or baseline, without other causes. Hematologic DLTs: Gr 4 neutropenia ≥7 days. Gr 4 thrombocytopenia. Gr 3 thrombocytopenia with bleeding or platelet transfusion. Febrile neutropenia. Gr 3 hemolysis requiring intervention. Gr 4 anemia not due to underlying disease. Dermatologic DLTs: Gr 4 rash. Gr 3 rash not improving to ≤Gr 1 after 1-2 week delay. Other DLTs: Gr 2-4 eye issues, Gr 3-4 toxicities, excluding specific Gr 3 events like nausea, fever.
Time Frame: From first dose (Day 1) and up to 6 weeks
Population: All Treated Participants. Pre-specified to be only collected for Part 1A, 1B, 1C and 2A arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1

4. Primary Outcome: Part 1A, 1B and 1C and 2A: Number of Participants With Grade 3/Grade 4 Laboratory Abnormalities
Description: Blood samples were collected to assess the abnormalities in laboratory parameters. The laboratory parameters were graded by Common Terminology Criteria for Adverse Events (CTCAE). Grade 3=Severe; Grade 4=Life-threatening.
Time Frame: From first dose (Day 1) till 100 days after last dose (Up to approximately 27 months)
Population: All treated participants with available laboratory abnormality results. Pre-specified to be only collected for Part 1A, 1B, 1C and 2A arms.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18
Participants
  HEMOGLOBIN (Grade 3) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 2
  PLATELET COUNT (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PLATELET COUNT (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LEUKOCYTES (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LEUKOCYTES (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEUTROPHILS (ABSOLUTE) (Grade 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  NEUTROPHILS (ABSOLUTE) (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  LYMPHOCYTES (ABSOLUTE) (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  LYMPHOCYTES (ABSOLUTE) (Grade 3) | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 0 | 2 | 1 | 2 | 1 | 2
  LYMPHOCYTES (ABSOLUTE) (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  LYMPHOCYTES (ABSOLUTE) (Grade 4) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT (Grade 3) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ABSOLUTE NEUTROPHIL COUNT (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  APTT (Grade 3): number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 7
  APTT (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  APTT (Grade 4): number analyzed (Participants) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 1 | 0 | 1 | 7
  APTT (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALKALINE PHOSPHATASE (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ALKALINE PHOSPHATASE (Grade 3) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 1 | 0 | 0 | 1
  ALKALINE PHOSPHATASE (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ALKALINE PHOSPHATASE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ASPARTATE AMINOTRANSFERASE (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ASPARTATE AMINOTRANSFERASE (Grade 3) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  ASPARTATE AMINOTRANSFERASE (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ASPARTATE AMINOTRANSFERASE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ALANINE AMINOTRANSFERASE (Grade 3) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  ALANINE AMINOTRANSFERASE (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ALANINE AMINOTRANSFERASE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  G-GLUTAMYL TRANSFERASE (Grade 3): number analyzed (Participants) | 0 | 0 | 3 | 2 | 5 | 3 | 14 | 2 | 3 | 3 | 2 | 3 | 11
  G-GLUTAMYL TRANSFERASE (Grade 3) | 0 | 0 | 1 | 0 | 2 | 0 | 7 | 0 | 1 | 2 | 0 | 1 | 3
  G-GLUTAMYL TRANSFERASE (Grade 4): number analyzed (Participants) | 0 | 0 | 3 | 2 | 5 | 3 | 14 | 2 | 3 | 3 | 2 | 3 | 11
  G-GLUTAMYL TRANSFERASE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  BILIRUBIN, TOTAL (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  BILIRUBIN, TOTAL (Grade 3) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
  BILIRUBIN, TOTAL (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  BILIRUBIN, TOTAL (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREATININE (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  CREATININE (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CREATININE (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  CREATININE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CALCIUM (Grade 3): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 7
  CALCIUM (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CALCIUM (Grade 4): number analyzed (Participants) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 7
  CALCIUM (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PHOSPHORUS (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  PHOSPHORUS (Grade 3) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PHOSPHORUS (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  PHOSPHORUS (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ALBUMIN (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ALBUMIN (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  ALBUMIN (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  ALBUMIN (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AMYLASE (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 4 | 16
  AMYLASE (Grade 3) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  AMYLASE (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 4 | 16
  AMYLASE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  LIPASE (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 4 | 16
  LIPASE (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2
  LIPASE (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 4 | 16
  LIPASE (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  URIC ACID (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  URIC ACID (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  URIC ACID (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  URIC ACID (Grade 4) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
  HYPERNATREMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERNATREMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERNATREMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERNATREMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPONATREMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPONATREMIA (Grade 3) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 4
  HYPONATREMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPONATREMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERKALEMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERKALEMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERKALEMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERKALEMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOKALEMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPOKALEMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOKALEMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPOKALEMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERCALCEMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERCALCEMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERCALCEMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERCALCEMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOCALCEMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPOCALCEMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOCALCEMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPOCALCEMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERMAGNESEMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERMAGNESEMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPERMAGNESEMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPERMAGNESEMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  HYPOMAGNESEMIA (Grade 3): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPOMAGNESEMIA (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  HYPOMAGNESEMIA (Grade 4): number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 17
  HYPOMAGNESEMIA (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2C: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with a confirmed Best overall response of Complete Response (CR) or Partial Response (PR) by RECIST v1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose (Day 1) and up to 24 weeks
Population: All Treated Participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 5
percentage of participants | 20.0 [0.5 to 71.6]

6. Primary Outcome: Part 2C: Duration of Response (DOR)
Description: DOR is defined for participants who have a confirmed CR or PR as the date from first documented CR or PR per RECIST v1.1 to the date of the documentation of disease progression or death due to any cause, whichever is earlier.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose (Day 1) and up to 24 weeks
Population: All Treated Participants. Participants with CR or PR were included in the analysis.
Measure: Median (Full Range); unit: months
Arm/Group | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1
months | NA [NA to NA] — Not estimated due to inadequate number of events.

7. Primary Outcome: Part 2C: Progression Free Survival Rate at Week 24
Description: Progression Free Survival Rates at 24 weeks is defined as the percentage of participants who achieve PFS at 24 weeks. PFS for a participant is defined as the time from randomization date to the date of first objectively documented disease progression by investigator per response evaluation criteria in solid tumors (RECIST) v1.1 or death due to any cause, whichever occurs first. Based on Kaplan-Meier Estimates.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum during the study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Week 24
Population: All Treated Participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 5
percentage of participants | 80.0 [20.4 to 96.9]

8. Secondary Outcome: Objective Response Rate (ORR)
Description: as for outcome 5
Time Frame: From first dose (Day 1) and up to 24 weeks
Population: All Treated Participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18
percentage of participants | 0.0 [0.0 to 97.5] | 0.0 [0.0 to 84.2] | 0.0 [0.0 to 70.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 16.8] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 60.2] | 22.2 [6.4 to 47.6] | 33.3 [4.3 to 77.7] | 5.6 [0.1 to 27.3]

9. Secondary Outcome: Duration of Response
Description: as for outcome 6
Time Frame: From first dose (Day 1) and up to 24 weeks
Population: All Treated Participants. Participants with CR or PR were included in the analysis.
Measure: Median (Full Range); unit: percentage of participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 1
percentage of participants |  |  |  |  |  |  |  |  |  |  | NA [NA to NA] — Not evaluable due to inadequate number of events | NA [NA to NA] — Not evaluable due to inadequate number of events | NA [NA to NA] — Not evaluable due to inadequate number of events

10. Secondary Outcome: Progression Free Survival Rate at Week 24
Description: as for outcome 7
Time Frame: Week 24
Population: All Treated Participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 66.7 [5.4 to 94.5] | 100.0 [100.0 to 100.0] | 75.0 [31.5 to 93.1] | 100.0 [100.0 to 100.0] | 70.0 [45.1 to 85.3] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 75.0 [12.8 to 96.1] | 93.3 [61.3 to 99.0] | 66.7 [19.5 to 90.4] | 61.1 [35.3 to 79.2]

11. Secondary Outcome: Maximum Observed Concentration (Cmax) of BMS-986207
Description: Cmax is defined as maximum plasma concentration of the drug.
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: All treated participants who have evaluable concentration-time data were included in the analysis. Only participants with evaluable concentration-time data at particular timepoint are considered in the analysis. Participant in Part 1A BMS-986207 Safety Run In did not meet criteria of evaluable concentration-time data hence not included in the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
ng/mL
  Cycle 1 Day 1 | 4952 (34) | 27291 (11) | 78548 (29) | 249112 (16) | 439192 (15) | 259914 (27) | 48703 (86) | 67136 (31) | 510696 (29) | 124997 (27) | 446640 (20) | 215247 (31) | 257979 (35)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 7540 (NA) — Not evaluable due to inadequate number of participants analyzed | 41200 (NA) — Not evaluable due to inadequate number of participants analyzed | 112632 (36) | 349009 (28) | 646106 (7) | 351683 (29) | 33291 (18) | 73100 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 486000 (NA) — Not evaluable due to inadequate number of participants analyzed | 165211 (20) | 442029 (41) | 272349 (65) | 322580 (40)

12. Secondary Outcome: BMS-986207 Time to Maximum Concentration (Tmax)
Description: Time to observed maximum concentration (Tmax) is defined as the amount of time in hours for a drug to reach the maximum concentration after administration.
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
hours
  Cycle 1 Day 1 | 2.20 (169) | 1.07 (9) | 1.00 (5) | 1.29 (59) | 1.59 (72) | 1.11 (31) | 9.63 (3383) | 0.962 (5) | 1.47 (75) | 1.63 (110) | 1.94 (50) | 1.53 (62) | 1.64 (23)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 5.00 (NA) — Not evaluable due to inadequate number of participants analyzed | 0.983 (NA) — Not evaluable due to inadequate number of participants analyzed | 0.989 (3) | 4.92 (515) | 10.0 (190) | 4.08 (291) | 2.51 (96) | 1.00 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 3.98 (NA) — Not evaluable due to inadequate number of participants analyzed | 1.88 (82) | 1.00 (0) | 1.03 (9) | 1.42 (37)

13. Secondary Outcome: BMS-986207 Area Under the Serum Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC (0-T))
Description: BMS-986207 area under the serum concentration-time curve from time zero to time of last quantifiable concentration (AUC (0-T)).
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
h*ng/mL
  Cycle 1 Day 1 | 903246 (16) | 4040645 (20) | 11778859 (27) | 39736190 (26) | 66647788 (15) | 33053505 (37) | 4954133 (63) | 7568790 (58) | 103780934 (21) | 26213882 (34) | 55152586 (79) | 34199336 (38) | 38608827 (34)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 1433844 (NA) — Not evaluable due to inadequate number of participants analyzed | 8631703 (NA) — Not evaluable due to inadequate number of participants analyzed | 21669222 (46) | 79172947 (31) | 151321351 (17) | 74976626 (45) | 5329459 (43) | 16061212 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 113248878 (NA) — Not evaluable due to inadequate number of participants analyzed | 42867360 (24) | 133901271 (49) | 56012897 (46) | 53257007 (82)

14. Secondary Outcome: BMS-986207 Area Under the Serum Concentration-time Curve in One Dosing Interval AUC (TAU)
Description: Blood samples were collected for assessing AUC (TAU).
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
h*ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 4 | 18 | 5
  Cycle 1 Day 1 | 903246 (16) | 4040645 (20) | 11778859 (27) | 42372351 (16) | 66647788 (15) | 36019071 (29) | 5436490 (49) | 7962140 (46) | 107854224 (27) | 27192752 (27) | 85887190 (28) | 35370530 (35) | 38608827 (34)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 1433844 (NA) — Not evaluable due to inadequate number of participants analyzed | 8631703 (NA) — Not evaluable due to inadequate number of participants analyzed | 21669222 (46) | 75841795 (35) | 151321351 (17) | 72506970 (42) | 6228807 (14) | 16061212 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 113248878 (NA) — Not evaluable due to inadequate number of participants analyzed | 44114081 (23) | 124674549 (38) | 56012897 (46) | 53257007 (82)

15. Secondary Outcome: BMS-986207 Observed Serum Concentration at the End of a Dosing Interval (Ctau)
Description: Blood samples were collected for assessing Ctau.
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 6 | 18 | 5
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 18 | 4 | 18 | 5
  Cycle 1 Day 1 | 1657 (24) | 6526 (41) | 20264 (34) | 79783 (18) | 118571 (29) | 51893 (53) | 5875 (31) | 9560 (158) | 66597 (44) | 17353 (56) | 75172 (36) | 26556 (54) | 22879 (61)
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 2790 (NA) — Not evaluable due to inadequate number of participants analyzed | 18500 (NA) — Not evaluable due to inadequate number of participants analyzed | 43315 (45) | 157016 (48) | 383682 (37) | 136133 (54) | 11449 (24) | 34400 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 83300 (NA) — Not evaluable due to inadequate number of participants analyzed | 34396 (43) | 149964 (23) | 61568 (53) | 37051 (272)

16. Secondary Outcome: BMS-986207 Total Body Clearance (CLT)
Description: Blood samples were collected for assessing CLT.
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 1 | 9 | 2 | 4 | 2
L/h
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 0.014 (NA) — Not evaluable due to inadequate number of participants analyzed | 0.009 (NA) — Not evaluable due to inadequate number of participants analyzed | 0.011 (46) | 0.011 (35) | 0.011 (17) | 0.011 (42) | 0.013 (14) | 0.015 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 0.014 (NA) — Not evaluable due to inadequate number of participants analyzed. | 0.011 (23) | 0.007 (13) | 0.011 (46) | 0.011 (82)

17. Secondary Outcome: BMS-986207 Average Concentration Over a Dosing Interval (Css-avg)
Description: Blood samples were collected for assessing Css-avg.
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 1 | 9 | 2 | 4 | 2
ng/mL
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 4281 (NA) — Not evaluable due to inadequate number of participants analyzed | 25746 (NA) — Not evaluable due to inadequate number of participants analyzed | 64581 (46) | 225882 (35) | 451954 (17) | 209969 (46) | 18650 (15) | 48112 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 168655 (NA) — Not evaluable due to inadequate number of participants analyzed | 67521 (23) | 247899 (37) | 113134 (46) | 103591 (78)

18. Secondary Outcome: BMS-986207 Ratio of an Exposure Measure at Steady State to That After the First Dose (AI_TAU)
Description: Blood samples were collected for assessing AI_TAU.
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 1 | 9 | 2 | 4 | 2
Ratio
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 3 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 1.42 (NA) — Not evaluable due to inadequate number of participants analyzed | 2.00 | 1.94 (17) | 1.91 (29) | 2.04 (2) | 1.97 (11) | 1.35 (57) | 1.93 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2 | 4 | 2
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 1.40 (NA) — Not evaluable due to inadequate number of participants analyzed | 1.47 (11) | 1.19 (34) | 1.46 (8) | 1.40 (102)

19. Secondary Outcome: BMS-986207 Effective Elimination Half-life That Explains the Degree of Accumulation Observed for a Specific Exposure Measure (T-HALFeff)
Description: Blood samples were collected for assessing T-HALFeff. Exposure measure includes AUC[TAU].
Time Frame: Day 1 of Cycle 1, Cycle 2 and Cycle 3 (Each cycle is of 8 weeks)
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 2 | 1 | 1 | 9 | 1 | 4 | 1
hours
  Cycle 1 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1: number analyzed (Participants) | 1 | 1 | 3 | 4 | 2 | 5 | 2 | 1 | 0 | 0 | 0 | 0 | 0
  Cycle 2 Day 1 | 189 (NA) — Not evaluable due to inadequate number of participants analyzed | 334 (NA) — Not evaluable due to inadequate number of participants analyzed | 319 (26) | 306 (43) | 344 (3) | 338 (14) | 293 (11) | 317 (NA) — Not evaluable due to inadequate number of participants analyzed |  |  |  |  |
  Cycle 3 Day 1: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 1 | 4 | 1
  Cycle 3 Day 1 |  |  |  |  |  |  |  |  | 372 (NA) — Not evaluable due to inadequate number of participants analyzed | 390 (32) | 317 (NA) — Not evaluable due to inadequate number of participants analyzed | 294 (16) | 722 (NA) — Not evaluable due to inadequate number of participants analyzed

20. Secondary Outcome: Number of Participants With Positive Anti-BMS-986207-Antibodies Results
Description: Participants who were treated with BMS-986207 and at least one post-baseline evaluable ADA assessment were considered in the analysis
Time Frame: From first dose (Day 1) till 100 days after last dose (Up to approximately 27 months)
Population: All Treated Participants with Baseline and at Least One Post-baseline Evaluable ADA Assessment were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
Number analyzed (Participants) | 1 | 2 | 3 | 4 | 8 | 4 | 20 | 4 | 4 | 4 | 14 | 2 | 5 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality was collected from randomization till death due to any cause (Up to approximately 85 months). Serious adverse events and non serious adverse events were collected from from first dose (Day 1) until 100 days after last dose (Up to approximately 27 months)
Description: All Cause Mortality , Serious and Others (Non-Serious) Adverse events were collected for All Treated Participants.
Arm/Group | Part 1A BMS-986207 Safety Run In | Part 1A BMS-986207 20 mg | Part 1A BMS-986207 80 mg | Part 1A BMS-986207 240 mg | Part 1A BMS-986207 800 mg | Part 1A BMS-986207 1600 mg | Part 2A BMS-986207 800 mg (CRC) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg | Part 1B BMS-986207 240 mg + Nivolumab 240 mg | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/2 | 3/3 | 2/4 | 5/8 | 2/4 | 15/20 | 2/4 | 4/4 | 4/4 | 7/18 | 3/6 | 13/18 | 3/5
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2 | 3/3 | 3/4 | 5/8 | 1/4 | 11/20 | 3/4 | 2/4 | 1/4 | 6/18 | 4/6 | 11/18 | 5/5
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2 | 3/3 | 4/4 | 8/8 | 4/4 | 20/20 | 3/4 | 4/4 | 4/4 | 18/18 | 6/6 | 18/18 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A BMS-986207 Safety Run In (N=1) | Part 1A BMS-986207 20 mg (N=2) | Part 1A BMS-986207 80 mg (N=3) | Part 1A BMS-986207 240 mg (N=4) | Part 1A BMS-986207 800 mg (N=8) | Part 1A BMS-986207 1600 mg (N=4) | Part 2A BMS-986207 800 mg (CRC) (N=20) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg (N=4) | Part 1B BMS-986207 240 mg + Nivolumab 240 mg (N=4) | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg (N=4) | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg (N=18) | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg (N=6) | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg (N=18) | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg (N=5)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Allergic oedema (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stoma site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 1 | 3 | 1 | 5 | 1 | 2 | 1 | 0 | 2 | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A BMS-986207 Safety Run In (N=1) | Part 1A BMS-986207 20 mg (N=2) | Part 1A BMS-986207 80 mg (N=3) | Part 1A BMS-986207 240 mg (N=4) | Part 1A BMS-986207 800 mg (N=8) | Part 1A BMS-986207 1600 mg (N=4) | Part 2A BMS-986207 800 mg (CRC) (N=20) | Part 1B BMS-986207 80 mg + Nivolumab 240 mg (N=4) | Part 1B BMS-986207 240 mg + Nivolumab 240 mg (N=4) | Part 1B BMS-986207 1600 mg + Nivolumab 480 mg (N=4) | Part 1B: BMS-986207 480 mg + Nivolumab 480 mg (N=18) | Part 1C BMS-986207 1200 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg (N=6) | Part 1C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg (N=18) | Part 2C BMS-986207 600 mg + Nivolumab 360 mg + Ipilimumab 1 mg/kg (N=5)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 2 | 3 | 3 | 3 | 4
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 0 | 5 | 1 | 0 | 0 | 1 | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Aptyalism (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 4 | 0 | 0 | 2 | 1 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 2 | 3 | 1 | 1 | 1 | 4 | 1 | 3 | 2
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagomediastinal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 3 | 1 | 0 | 1 | 2 | 0 | 2 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 5 | 1 | 4 | 0 | 1 | 2 | 5 | 0 | 5 | 3
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nodule (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 3 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 0 | 2 | 2 | 2 | 0 | 7 | 1
Swelling face (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vessel puncture site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cryptosporidiosis infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Encephalitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Stoma site abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stoma site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adjusted calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 1
Ammonia increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 3 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 2
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Blood calcium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 2
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Blood potassium decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood sodium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood urea increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Drug level increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 2
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 2 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 2 | 2 | 1 | 5 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3 | 1 | 4 | 1 | 0 | 1 | 4 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 6 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Laryngeal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Drooling (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ulnar nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urogenital fistula (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 4 | 0 | 2 | 0 | 3 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 0 | 3 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 1 | 2 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 8 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/13/NCT02913313/Prot_SAP_000.pdf